CLINICAL TRIAL: NCT02910323
Title: The Will Erwin Headache Research Center Study of Cluster Headache and Trigeminal Neuralgia
Brief Title: The Will Erwin Headache Research Center - Cluster Headache Study
Acronym: WEC1
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mark J Burish, Assistant Professor, Neurosurgery, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0780
Record Dates: First submitted 2016-09-15; First posted 2016-09-22 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cluster Headache; Cluster Headaches and Other Trigeminal Autonomic Cephalgias; Paroxysmal Hemicrania; SUNCT; Hemicrania Continua; Trigeminal Neuralgia
MeSH Terms: conditions — Cluster Headache; Paroxysmal Hemicrania; Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, saliva, skin cells, other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental group: Patients with a history of Cluster Headaches and other TACs, or Trigeminal Neuralgia.
- Family/Healthy Controls: Healthy volunteer controls and family members may be enrolled for identification of genetic mutations.

SUMMARY:
The Will Erwin Headache Research Center Study of Cluster Headache and Trigeminal Neuralgia is a prospective, multicenter, observational research network for subjects with Cluster Headache and/or Trigeminal Neuralgia.

DETAILED DESCRIPTION:
The Will Erwin Headache Research Center will assemble a national registry of Cluster Headache patients and will sub-categorize and organize this cohort based on individuating characteristics including but not limited to type and severity of condition, associated symptoms, and medical/psychological issues (e.g., depression, disability, sleep). Detailed evaluations and classification will be completed for each enrolled subject. This will encompass genomic and epigenomic studies, past medical history, imaging reports, and specific physical exam results for each patient. It will also enable the study investigators to match patients with suitable interventional clinical trials.

Similar diseases, such as other paroxysmal hemicrania, SUNCT, SUNA, hemicrania continua, and trigeminal neuralgia may also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a trigeminal autonomic cephalalgia according to the International Headache Classification including episodic cluster headache, chronic cluster headache, episodic paroxysmal hemicrania, chronic paroxysmal hemicrania, episodic short-lasting unilateral neuralgiform headache attacks with conjunctival injection and tearing (SUNCT), chronic SUNCT, episodic short-lasting unilateral neuralgiform headache attacks with cranial autonomic symptoms (SUNA), chronic SUNA, and hemicrania continua. OR Diagnosis of a trigeminal neuralgia according to the International Headache Classification, including classical trigeminal neuralgia and symptomatic trigeminal neuralgia.
* Able to provide HIPAA authorization to share prior medical records/imaging.

Exclusion Criteria:

* Life expectancy less than 1 year, co-existing disease or other characteristic that precludes appropriate diagnosis of a trigeminal autonomic cephalalgia or trigeminal neuralgia.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Inability or unwillingness of subject or legal guardian/representative to give informed consent.

Inclusion Criteria for Healthy Volunteers:

* Inclusion criteria is willingness to consent and be of age 18 and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cluster Headache and Trigeminal Neuralgia patients, family members and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-05; Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
HIT-6 scale | Through study completion, an average of 5 years
Morningness-eveningness scale | Through study completion, an average of 5 years
GAD-7 scale | Through study completion, an average of 5 years

SECONDARY OUTCOMES:
Genetic markers | Through study completion, an average of 5 years
  Results of GWAS or other genetic tests
Molecular biomarkers | Through study completion, an average of 5 years
  Results of ELISAs for autonomic, hypothalamic, and pain signalling molecules

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burish, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276